CLINICAL TRIAL: NCT02313675
Title: Comparing Pain Outcomes of Intra-operative IV Tylenol and/or IV Toradol Administration for Carpal Tunnel Release and Distal Radius Fracture Surgeries
Brief Title: Pain Outcomes of Intra-operative IV Tylenol and/or IV Toradol for Carpal Tunnel and Distal Radius Fracture Surgeries
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: John Fowler (Other)
Responsible Party: Sponsor-Investigator, John Fowler, MD, University of Pittsburgh
Organization: University of Pittsburgh (Other)
Allocation: Randomized | Model: Factorial | Masking: Triple | Purpose: Treatment
Other Study IDs: PRO14110464
Record Dates: First submitted 2014-12-08; First posted 2014-12-10 (Estimated); Results first posted 2018-05-04 (Actual); Last update posted 2018-05-04 (Actual); Status verified 2018-04

CONDITIONS: Postoperative Pain; Carpal Tunnel Release; Distal Radius Fracture
Keywords: carpal tunnel syndrome; opioid analgesics; postoperative pain; IV tylenol; IV toradol
MeSH Terms: conditions — Pain, Postoperative; Wrist Fractures; Carpal Tunnel Syndrome | interventions — Acetaminophen; Ketorolac Tromethamine; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- IV tylenol (Experimental): One time intra-operative IV acetaminophen administration
  Interventions: Drug: Acetaminophen
- IV toradol (Experimental): One time intra-operative IV ketorolac thromethamine administration
  Interventions: Drug: Ketorolac Tromethamine
- IV tylenol/toradol combination (Experimental): One time intra-operative IV combination of acetaminophen/ketorolac administration
  Interventions: Drug: Acetaminophen; Drug: Ketorolac Tromethamine
- saline (Placebo Comparator): One time intra-operative 50ml IV normal saline administration
  Interventions: Drug: Saline

INTERVENTIONS:
Drug: Acetaminophen
  Other Names: tylenol
  Arms: IV tylenol; IV tylenol/toradol combination
Drug: Ketorolac Tromethamine
  Other Names: toradol
  Arms: IV toradol; IV tylenol/toradol combination
Drug: Saline
  Arms: saline

SUMMARY:
The purpose of this study is to determine the efficacy of intra-operative administration of IV tylenol and/or IV toradol in minimizing post-operative pain for carpal tunnel patients and distal radius fracture patients.

DETAILED DESCRIPTION:
The study population will include patients presenting for surgery with carpal tunnel syndrome as well as surgical treatment of distal radius fracture. Patients will be treated intra-operatively with either IV tylenol, IV toradol, both, or neither. All patients will receive the standard post-operative prescriptions for pain management. Daily pain surveys scoring pain from 0-10 will be distributed to the subjects to be filled out over the course of 10 days prior to first post-operative visit, usually 10-14 days later. Number of pain pills used before the first post-operative visit will also be measured.

We hypothesize that the effects of intra-operative administration of IV tylenol and/or IV toradol will have a significant effect on decreasing post-operative pain in the first 10 days following distal radius fracture surgeries, with a significant difference in pain described as at least a 2 points on a 0-10 pain scale.

We also hypothesize that intra-operative administration of IV tylenol and/or IV toradol will not have such significant effect on decreasing post-operative pain for carpal tunnel release surgery.

A secondary aim is to evaluate the post-operative opioid consumption of patients within these treatment groups. We hypothesize that opioid consumption will be decreased in the groups receiving IV tylenol and/or toradol for distal radius fracture surgery compared to the placebo group. We do not expect such a difference for the carpal tunnel release surgery group.

ELIGIBILITY:
Inclusion Criteria:

* carpal tunnel release surgery candidates,
* distal radius fracture surgery candidates

Exclusion Criteria:

* under 18 years of age,
* pregnant women,
* prisoners

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2015-05; Primary Completion 2017-05-01 (Actual); Study Completion 2017-05-01 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Kaufmann Building, Pittsburgh, Pennsylvania, United States

REFERENCES:
- [Background] Hahn TW, Mogensen T, Lund C, Jacobsen LS, Hjortsoe NC, Rasmussen SN, Rasmussen M. Analgesic effect of i.v. paracetamol: possible ceiling effect of paracetamol in postoperative pain. Acta Anaesthesiol Scand. 2003 Feb;47(2):138-45. doi: 10.1034/j.1399-6576.2003.00046.x. PMID 12631041
- [Background] Baley K, Michalov K, Kossick MA, McDowell M. Intravenous acetaminophen and intravenous ketorolac for management of pediatric surgical pain: a literature review. AANA J. 2014 Feb;82(1):53-64. PMID 24654353
- [Background] Smith HS. Perioperative intravenous acetaminophen and NSAIDs. Pain Med. 2011 Jun;12(6):961-81. doi: 10.1111/j.1526-4637.2011.01141.x. Epub 2011 May 31. PMID 21627768
- [Background] Alhashemi JA, Daghistani MF. Effects of intraoperative i.v. acetaminophen vs i.m. meperidine on post-tonsillectomy pain in children. Br J Anaesth. 2006 Jun;96(6):790-5. doi: 10.1093/bja/ael084. Epub 2006 Apr 13. PMID 16613928

RESULTS

PARTICIPANT FLOW:
Groups:
- IV Tylenol: One time intra-operative IV acetaminophen administration
  Acetaminophen
- IV Toradol: One time intra-operative IV ketorolac thromethamine administration
  Ketorolac Tromethamine
- IV Tylenol/Toradol Combination: One time intra-operative IV combination of acetaminophen/ketorolac administration
  Acetaminophen
  Ketorolac Tromethamine
- Saline: One time intra-operative 50ml IV normal saline administration
  Saline
Period: Overall Study
Arm/Group | IV Tylenol | IV Toradol | IV Tylenol/Toradol Combination | Saline
Started | 11 | 11 | 11 | 11
Completed | 11 | 11 | 11 | 11
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | IV Tylenol | IV Toradol | IV Tylenol/Toradol Combination | Saline | Total
Number analyzed (Participants) | 11 | 11 | 11 | 11 | 44
Age, Continuous [Mean (Full Range); unit: years] | 57 [48 to 67] | 48 [37 to 58] | 43 [32 to 53] | 55 [45 to 65] | 51 [43 to 63]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 8 | 6 | 6 | 28
  Male | 3 | 3 | 5 | 5 | 16
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Postoperative Pain (Pain Scores From 0-10 Scale)
Description: This is an ordinal pain scale. The patient picks a number from 0-10 scale every 4 hours for 7 days post-operatively. 0 is no pain, 10 is the worst pain imaginable. Lower scores would be preferable to higher scores.
Time Frame: 7 days
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | IV Tylenol | IV Toradol | IV Tylenol/Toradol Combination | Saline
Number analyzed (Participants) | 11 | 11 | 11 | 11
units on a scale | 2.0 [1.7 to 2.3] | 2.9 [2.6 to 3.2] | 2.7 [2.3 to 3.0] | 2.0 [1.7 to 2.3]

2. Secondary Outcome: Opioid Consumption (Number of Pills Taken)
Description: Daily opioid consumption assessed as number of pills taken that day, each day for 7 days post-operatively
  Outcome measure reported below is mean number of opioid pills consumed per day.
Time Frame: 7 days
Measure: Mean (Full Range); unit: pills consumed
Arm/Group | IV Tylenol | IV Toradol | IV Tylenol/Toradol Combination | Saline
Number analyzed (Participants) | 11 | 11 | 11 | 11
pills consumed | 0.2 [0 to 12] | 0.7 [0 to 16] | 1.0 [0 to 20] | 0.7 [0 to 16]

ADVERSE EVENTS:
Time Frame: Time frame is 90 days after surgery
Arm/Group | IV Tylenol | IV Toradol | IV Tylenol/Toradol Combination | Saline
All-Cause Mortality (participants affected / at risk) | 0/11 | 0/11 | 0/11 | 0/11
Serious Adverse Events (participants affected / at risk) | 0/11 | 0/11 | 0/11 | 0/11
Other Adverse Events (participants affected / at risk) | 0/11 | 0/11 | 0/11 | 0/11

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2017-01-25): https://cdn.clinicaltrials.gov/large-docs/75/NCT02313675/Prot_000.pdf
  • Statistical Analysis Plan (2017-01-25): https://cdn.clinicaltrials.gov/large-docs/75/NCT02313675/SAP_001.pdf